CLINICAL TRIAL: NCT04693052
Title: Attitudes Towards Receiving Mental Health Care Using Telehealth During the COVID-19 Pandemic
Brief Title: Attitudes Towards Receiving Mental Health Care Using Telehealth During the Coronavirus Disease 2019 (COVID-19) Pandemic
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: STU00213696
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psychiatric Disorder; Mental Health Disorder; Stress; Adjustment Disorders
Keywords: Telehealth; Telemedicine; Telepsych; Telepsychiatry; Telepsychology; Telemental health; Survey; Attitudes; COVID-19; pandemic; mental health; therapy; psychiatry
MeSH Terms: conditions — Mental Disorders; Adjustment Disorders; Behavior; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mental Health patients starting pre-COVID: Patients receiving mental health care prior to and during the COVID-19 pandemic
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — This is a self-reported survey study about receiving mental health care during the COVID-19 pandemic

SUMMARY:
The purpose of this study is to collect patients' experiences and feedback to better understand and improve mental health care using telehealth services. This is critically important as telehealth appointments, including both phone and video calls, continue to be offered for regular appointments to reduce in-person interaction as a preventive measure to help control the spread of COVID-19.

DETAILED DESCRIPTION:
Studying patients' perceived benefits and challenges of using telehealth services for mental health care will allow us to prioritize improvements to the telehealth experience and potentially, patient adoption of and comfort with remote appointments. This study's results would also inform policy makers and insurance companies about the potential utility of delivering mental health care through telehealth, even beyond the duration of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and over who received mental health care through Northwestern prior to telehealth implementation from March 15th 2019 to March 14th 2020, and had at least one mental health care appointment through Northwestern between March 15th 2020 and September 30th 2020.

Exclusion Criteria:

* Adults unable to access study questionnaires via computer or mobile device

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People receiving mental health care at Northwestern Medicine during the COVID-19 pandemic
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rado, MD, Principal Investigator — Northwestern University
Locations (1):
- Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic: No interventions: This is a self-reported survey study about receiving mental health care during the coronavirus disease 2019 (COVID-19) pandemic
Period: Overall Study
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic
Started | 605
Completed | 605
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic: No interventions: This is a self-reported survey study about receiving mental health care during the COVID-19 pandemic
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic
Number analyzed (Participants) | 605
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 participants with no telehealth use were excluded Remaining difference because some participants did not respond to demographic questions. Questions were not mandatory
  Participants
    number analyzed (Participants) | 600
    <=18 years | 0
    Between 18 and 65 years | 459
    >=65 years | 141
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 participants excluded because they did not use telehealth Remaining difference because some participants did not respond to demographic questions. Questions were not mandatory
  Participants
    number analyzed (Participants) | 597
    Female | 418
    Male | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants excluded because they did not use telehealth
  Participants
    number analyzed (Participants) | 602
    Hispanic or Latino | 55
    Not Hispanic or Latino | 494
    Unknown or Not Reported | 53
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants excluded because they did not use telehealth
  Participants
    number analyzed (Participants) | 602
    American Indian or Alaska Native | 13
    Asian | 31
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 84
    White | 457
    More than one race | 0
    Unknown or Not Reported | 17
Household income [Count of Participants; unit: Participants] — Population: 3 participants excluded due to not using telehealth Some patients did not respond to question
  Participants
    number analyzed (Participants) | 597
    Prefer not to answer | 80
    <10k | 50
    10K - <15k | 37
    15K - <30k | 64
    30K - <50k | 62
    50K - <75k | 84
    75K - <100k | 51
    100K - <200k | 122
    >200k | 47

OUTCOME MEASURES:

1. Primary Outcome: Patient Choosing Telehealth as an Option for Future Care
Description: Patients choosing telehealth or not for future case, or unsure)
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Groups:
- Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic Using Telehealth: No interventions: This is a self-reported survey study about receiving mental health care during the COVID-19 pandemic
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic Using Telehealth
Number analyzed (Participants) | 602
Participants
  Yes | 523
  No | 43
  Unsure | 36

2. Primary Outcome: Comparison Between In-person and Telehealth
Description: Subjects will reply on a 5 point scale (Telehealth much better, Telehealth better, about the same, In-person better, In-person much better
  Items compared: Quality of mental health care, ability to express one self, time & money savings, ease of managing responsibilities, length of wait times and appointments missed
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic
Number analyzed (Participants) | 598
Participants
  Telehealth much better | 53
  Telhealth better | 43
  About the same | 335
  In-person better | 115
  In-person much better | 52

3. Primary Outcome: Patient Satisfaction With Telehealth
Description: Subjects will reply on a 5 point scale (Extremely satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, Extremely Dissatisfied)
  No standard questionnaire. Internally developed questions
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic Using Telehealth
Number analyzed (Participants) | 598
Participants
  Extremely satisfied | 278
  Satisfied | 227
  Neither satisfied nor dissatisfied | 56
  Unsatisfied | 30
  Extremely unsatisfied | 7

4. Primary Outcome: Patient Comfort Using Telehealth
Description: Subjects will reply on a 5 point scale (Extremely comfortable, Comfortable, Neither comfortable nor uncomfortable, Uncomfortable, Extremely uncomfortable)
  No standard questionnaire. Internally developed questions
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic Using Telehealth
Number analyzed (Participants) | 596
Participants
  Extremely Comfortable | 297
  Comfortable | 234
  Neither comfortable nor uncomfortable | 36
  Uncomfortable | 22
  Extremely uncomfortable | 7

5. Primary Outcome: Patient Easy of Using Telehealth
Description: Subjects will reply on a 5 point scale (Extremely easy, Easy, Neither easy nor difficult, Difficult, Extremely difficult)
  No standard questionnaire. Internally developed questions
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic
Number analyzed (Participants) | 595
Participants
  Extremely easy | 318
  Easy | 209
  Neither easy nor difficult | 48
  Difficult | 16
  Extremely difficult | 4

ADVERSE EVENTS:
Description: not applicable. This was a one-point-in-time survey study. Adverse events were not assessed.
Arm/Group | Patients Receiving Mental Health Care Prior to and During the COVID-19 Pandemic
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT04693052/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT04693052/SAP_001.pdf